CLINICAL TRIAL: NCT07317427
Title: Clinical Study for Precise Image for Interventional CT for Incisive CT and CT 5300 Systems
Brief Title: Precise Image for Interventional CT
Status: Not yet recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Philips Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Precise Image for CCT
Record Dates: First submitted 2025-09-23; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
The purpose of this clinical study is to assess the performance of the Precise Image reconstruction algorithm on interventional CT images acquired from adult patients (>18 years old). The analysis will focus on the performance of Precise Image for scans in which procedural instruments (e.g., needle, probe, screw) are present. Clinical data generated from this study is intended to support a proposed expansion of the Indications for Use of Precise Image.

The study has two objectives:

1. To evaluate the image quality for procedural guidance and procedural confidence of Precise Image compared to the standard-of-care reference (iDose4) for:

   * Interventional CT images of adult patients (>18 years old).
2. To demonstrate non-inferiority of Precise Image to iDose4 for the relevant interventional CT images.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scanned by FDA-cleared and marketed Philips Incisive CT or CT 5300 systems, and according to the department standard of care clinical protocols for the applicable clinical scans.
* Subject age: >18 years old.
* Presence of procedural instrument(s) (e.g., needle, probe, screw) in the CT images.

Exclusion Criteria:

* Subject age: 18 years old and below.
* Absence of procedural instrument(s) (e.g., needle, probe, screw) in the CT images.
* Scans that were acquired using a kilovoltage peak of 70 kVp (as Precise Image does not support a kilovoltage peak lower than 80 kVp).
* Scans that the site interventional radiologists have deemed non-suitable for procedural guidance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the CT image quality of Precise Image reconstructions via a 5-point Likert Scale | Reading session at 4 months
  The image quality of Precise Image reconstructions is non-inferior to iDose4 reconstructions for interventional CT images of adult patients. Measurement will be done via 5-point Likert Scale for Image Quality where 5 is excellent and 1 is poor image quality.